CLINICAL TRIAL: NCT01958216
Title: In Vivo TICE (TransIntestinal Cholesterol Excretion) Measurement in Bile Duct Diverted Patients
Brief Title: in Vivo TICE (TransIntestinal Cholesterol Excretion)
Acronym: in vivoTICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RC11_0008
Record Dates: First submitted 2013-09-30; First posted 2013-10-09 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-09

CONDITIONS: Occlusion of Bile Duct With an External Bile Diversion.
Keywords: TICE-human-stable isotopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Trans-intestinal cholesterol excretion in vivo (Other): Measuring trans-intestinal cholesterol excretion in vivo in bile diverted patients
  Interventions: Other: Intravenous injection of deuterated cholesterol diluted in intralipid 20%

INTERVENTIONS:
Other: Intravenous injection of deuterated cholesterol diluted in intralipid 20% — At day 0, bile diverted patients will receive an intravenous injection of deuterated cholesterol diluted in intralipid 20%. The plasma, biliary and fecal content of deuterated cholesterol will be measured, by mass spectrometry, at 24, 48 and 72 hours after the initial input.

SUMMARY:
So far, the liver has been the main target for cholesterol elimination. However, several recent studies performed in mice have described a new route of cholesterol excretion, the Trans-Intestinal Cholesterol Excretion or TICE. TICE allows direct elimination of plasma cholesterol in the feces directly via the intestine. Until now, only indirect evidence suggests that TICE is also active in humans, the goal of this proof of concept study is to provide the first proof of its existence in humans by using stable isotopes in patients with bile duct diversion.

ELIGIBILITY:
Inclusion Criteria:

- External bile duct diverted patients

Exclusion Criteria:

* Inflammatory bowel disease
* Aphagia
* Renal or hepatocellular insufficiency
* Primary intestinal tumor
* Cholangitis or severe sepsis
* Acute or chronic diarrhea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Measuring trans-intestinal cholesterol excretion in vivo in bile diverted patients | Day 3
  Measuring trans-intestinal cholesterol excretion in vivo in bile diverted patients

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Cariou, Pofessor, Principal Investigator — Nantes University Hospital
Locations (1):
- University Hospital, Nantes, France

REFERENCES:
- [Derived] Moreau F, Blanchard C, Perret C, Flet L, Douane F, Frampas E, Mirallie E, Croyal M, Aguesse A, Krempf M, Prieur X, Pichelin M, Cariou B, Le May C. In vivo evidence for transintestinal cholesterol efflux in patients with complete common bile duct obstruction. J Clin Lipidol. 2019 Jan-Feb;13(1):213-217.e1. doi: 10.1016/j.jacl.2018.09.010. Epub 2018 Sep 21. PMID 30342919